CLINICAL TRIAL: NCT07159243
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Parallel-designed Clinical Study to Evaluate the Efficacy and Safety of HL-1186 in Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: Evaluate the Efficacy and Safety of HL-1186 in Patients With Diabetic Peripheral Neuropathic Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PY-HL-1186-II-01
Record Dates: First submitted 2025-08-12; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HL-1186 Group 1 (Experimental): Each participant will receive HL-1186 for 12 weeks.
  Interventions: Drug: HL-1186
- HL-1186 Group 2 (Experimental): Each participant will receive HL-1186 for 12 weeks.
  Interventions: Drug: HL-1186
- HL-1186 Placebo (Placebo Comparator): Each participant will receive a matching placebo for 12 weeks.
  Interventions: Drug: HL-1186 placebo

INTERVENTIONS:
Drug: HL-1186 — HL-1186 tablet for oral administration.
  Arms: HL-1186 Group 1
Drug: HL-1186 — HL-1186 tablet for oral administration.
  Arms: HL-1186 Group 2
Drug: HL-1186 placebo — HL-1186 placebo tablet for oral administration.
  Arms: HL-1186 Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study design evaluating the safety, efficacy, and PK parameter of HL-1186 tablet for diabetic peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old (inclusive), regardless of gender.
2. With Type 1 or Type 2 diabetes mellitus, with a diagnosis of DPNP for at least 6 months.
3. Screening period: ADPS ranging from 4 to 9 points, and Visual Analog Scale (VAS) scores of 40mm - 90mm in two different days.
4. The hypoglycemic regimen has been stable for at least 4 weeks before enrollment, and the glycated hemoglobin (HbA1c) during the screening period is ≤ 9%.
5. Participants fully understand the purpose, characteristics, methods of the trial and possible adverse events, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Participants with any pain other than DPNP, or with other diseases that the investigator deems may affect the evaluation of DPNP.
2. Participants who are allergic to the active ingredients or excipients of HL-1186, HL-1186 placebo, or paracetamol tablets, or who have an allergic constitution, or have a history of allergies to ≥ 3 substances.
3. Participants who have used drugs that may damage nerves (such as tumor chemotherapy drugs) after being diagnosed with DPNP.
4. Participants who used any prohibited drugs within 2 weeks before screening (or within 5 half-lives after the last use of such prohibited drugs at the time of screening, whichever is longer).
5. Participants who had acute diabetic complications within 6 months before screening, such as diabetic ketoacidosis, hyperglycemic hyperosmolar state, lactic acidosis, acute severe hypoglycemia, etc., or had lower limb amputation (except toe amputation) at the time of screening.
6. Participants with clinically significant abnormalities in the 12-lead electrocardiogram (ECG) during the screening period (such as QTcF ≥ 450ms), or with severe cardiopulmonary diseases that the investigator deems inappropriate for inclusion, such as unstable angina pectoris, myocardial infarction, severe arrhythmias requiring treatment (such as grade Ⅲ atrioventricular block), NYHA cardiac function class ≥ Ⅲ, poorly controlled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg), recurrent asthma, etc.
7. Participants with neuropsychiatric system diseases that the investigator deems may affect the participant's evaluation of DPNP or scale evaluation, such as depression, anxiety, epilepsy, recurrent dizziness, memory and cognitive impairment, a history of suicide attempts or suicidal tendencies, etc.
8. Participants with a history of malignant tumors within 2 years before screening (except for participants with basal cell carcinoma, squamous cell carcinoma, and stage 0 cervical carcinoma in situ that have been confirmed cured by the investigator).
9. Participants with clinically significant and unstable diseases of the nervous system, mental system, ophthalmology, hepatobiliary system, respiratory system, hematological system, or cardiovascular system within 1 year before screening, and the investigator assesses that such diseases may endanger the participant's safety during the trial, restrict the participant from completing the study procedures, or affect the research purpose.
10. Participants with positive human immunodeficiency virus antibody, positive syphilis serological test, positive hepatitis B virus surface antigen with hepatitis B virus DNA > ULN, or positive hepatitis C virus antibody with hepatitis C virus RNA > ULN.
11. Participants with a history of alcoholism or drug abuse within 2 years before screening.
12. Female participants who are pregnant, breastfeeding (within 1 year after delivery), or with a positive pregnancy test.
13. Participants of childbearing potential who have plans to conceive, freeze or donate sperm/eggs from the time of signing the informed consent form until 6 months after the last dose, or who refuse to adopt effective contraceptive measures (complete abstinence, barrier methods, contraceptives, intrauterine devices, or having undergone sterilization surgery).
14. Participants who have participated in other drug or medical device trials within 3 months before screening or are currently participating in other clinical trials.
15. Participants deemed by the investigator to be unsuitable for participating in this study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in average daily pain score (ADPS) from baseline after 12 weeks of administration | From baseline to the end of treatment at 12 weeks
  Change from baseline in the weekly mean of the daily Numeric Pain Rating Scale (NPRS) score assessing the worst pain intensity in the last 24 hours. Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From first day of administration to the end of the last follow-up at Week 16

IPD SHARING:
Plan to Share IPD: No